CLINICAL TRIAL: NCT03203850
Title: A Phase II, Multicenter, Open-label, Randomized Two-year Study to Evaluate the Efficacy and Safety of Deferasirox Film-coated Tablet Versus Phlebotomy in Patients With Hereditary Hemochromatosis.
Brief Title: Study to Evaluate the Efficacy and Safety of Deferasirox Film-coated Tablet Versus Phlebotomy in Patients With Hereditary Hemochromatosis (HH)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to enrolment challenge
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CICL670F2203; 2016-002529-12 (EudraCT Number)
Record Dates: First submitted 2017-06-22; First posted 2017-06-29 (Actual); Results first posted 2024-06-07 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-05

CONDITIONS: Hereditary Hemochromatosis
Keywords: hereditary hemochromatosis; ICL670; deferasirox FCT; iron overload
MeSH Terms: conditions — Hemochromatosis; Iron Overload | interventions — Deferasirox; Phlebotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Deferasirox FCT Arm (Experimental): An initial dose of deferasirox FCT 7 mg/kg/day was used for 3 months (12 weeks), then was adjusted according to the serum ferritin (SF) level. Deferasirox was interrupted when the study-defined target SF ≤ 100 μg/L was achieved. Deferasirox was to be reinitiated when SF ≥ 300 μg/L, according to deferasirox label.
  Interventions: Drug: Deferasirox FCT
- phlebotomy (Active Comparator): Phlebotomy was conducted at a frequency determined by the physician. Phlebotomy was interrupted when the study-defined target SF ≤ 100 μg/L was achieved. Phlebotomy was to be reinitiated when SF > 100 μg/L, based on standard of care practice.
  Interventions: Procedure: Phlebotomy

INTERVENTIONS:
Drug: Deferasirox FCT — Taken orally once per day (QD) as a film coated tablet (FCT)
  Other Names: ICL670
  Arms: Deferasirox FCT Arm
Procedure: Phlebotomy — according to investigator's decision
  Arms: phlebotomy

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of deferasirox film coated tablet (FCT) versus phlebotomy for the management of iron overload in adults with Hereditary Hemochromatosis (HH) at risk of iron-related morbidity. This evaluation provided information on the two treatment options in terms of the rate of response of proportion of patients reaching the study target SF ≤ 100 μg/L and their associated safety profiles.

In addition to exploring the safety and efficacy of deferasirox FCT in hereditary hemochromatosis (HH), this study is being conducted to fulfill an FDA post-marketing requirement [PMC 750-10 (Exjade) /PMR 2888-8 (Jadenu)] to provide additional randomized data to confirm the ocular safety profile of deferasirox through detailed ocular assessments in patients treated with deferasirox FCT for 2 years.

DETAILED DESCRIPTION:
This was a Phase II, multicenter, open-label, randomized two-year study in adults with Hereditary Hemochromatosis (HH) confirmed by HH genotype with iron overload. Eligible subjects were identified during a 4-week screening period, then randomized in a 2:1 ratio to be treated with deferasirox FCT or phlebotomy for up to 24 months (104 weeks).

ELIGIBILITY:
Inclusion Criteria:

Written informed consent must be obtained prior to any screening procedures.

Patients eligible for inclusion must meet all following criteria prior to receiving study treatment:

1. Male or female ≥ 18-years-old 2. Documented genotype testing confirming homozygous for the C282Y mutation (C282Y/C282Y) 3. Transferrin saturation ≥ 45% (at either screening visit) 4. Serum ferritin (SF) ≥ 500 μg/L (at either screening visit)

-

Exclusion Criteria:

1. Medical conditions that preclude inclusion:

   * Iron overload not due to HH
   * Condition which might significantly alter the absorption, distribution, metabolism or excretion of oral deferasirox
   * Systemic disease which prevents taking study treatment or any contraindication to phlebotomy
   * Inflammatory condition or immunological disease which may interfere with the SF interpretation, such as an active infection, collagen vascular disorders, irritable bowel syndrome, lupus, or immune thrombocytopenia
   * Significantly impaired gastrointestinal function or disease that may significantly alter the absorption of oral deferasirox, e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection.
   * Psychiatric or addictive disorder which prevent giving informed consent or undergoing any of the treatment options or unwilling or unable to comply with the protocol
   * Uncontrolled or significant cardiac disease or symptomatic cardiac arrhythmias, e.g., sustained ventricular tachycardia and clinically significant second or third degree AV block without a pacemaker.
   * Illicit drug use and/or alcohol use, defined as an average alcohol consumption greater than one standard drink a day for women or two standard drinks a day for men within the 12 months prior to enrolment. A standard drink is generally considered to be 12 ounces of beer, 5 ounces of wine, or 1.5 ounces of 80-proof distilled spirits
   * Cirrhosis, including Child-Pugh class A, B, and C, diagnosed by liver biopsy, elastography, radiologic exams, or clinical criteria
   * Active hepatitis B or C (hepatitis B carrier will be allowed)
   * History of HIV seropositivity (ELISA or Western blot)
   * Organ transplant recipient
   * Malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, except localized basal cell carcinoma of the skin, or any history of hepatocellular carcinoma
2. Concomitant therapy that precludes enrollment:

   * Prior iron chelation therapy
   * Prohibited concomitant medications with deferasirox
3. Abnormal Laboratory Values:

   * Significant anemia that contraindicates phlebotomy (males with hemoglobin < 130g/L, females with hemoglobin < 120g/L) in both screening visit samples
   * Platelets ≤ 50 x 109/L in both screening visit samples
   * Urine protein/urine creatinine ratio > 1.0 mg/mg in both non-first void urine screening visit samples
   * Creatinine clearance ≤ 40 ml/min, or use the locally approved contraindication limit in prescribing information if it is stricter, in both screening visit samples
   * Serum creatinine > 1.5 x ULN in both screening visit samples
   * ALT ≥ 5 x ULN in both screening visit samples
   * Total bilirubin > 1.5 x ULN in both screening visit samples
4. Participation in an investigational study:

   * Observational registry study is allowable
   * Within 30 days prior to enrollment or within 5-half-lives of an investigational product, whichever is longer
   * Treatment with a systemic investigational drug within 4 weeks or topical investigational drug within 7 days of starting the study
5. Pregnancy and contraception:

   * Pregnant or nursing (lactating) women
   * Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless using basic methods of contraception, such as:
   * Total abstinence Periodic abstinence (calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are unacceptable methods.
   * Female sterilization (bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. If oophorectomy alone, hormone levels must confirm menopause.
   * Male sterilization (at least 6 months prior to screening). The vasectomized male must be the sole partner.
   * Barrier methods of contraception: condom or occlusive cap For UK: spermicidal foam/gel/film/cream/vaginal suppository
   * Placement of an intrauterine device or intrauterine system
   * Women considered as post-menopausal and not of childbearing potential are allowed to be enrolled in the trial if they have had 12 months of natural (spontaneous) amenorrhea with an expected clinical profile, e.g., age appropriate and history of vasomotor symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- Novartis Investigative Site, Leuven, Belgium
- France (2):
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Rennes
- Novartis Investigative Site, Sibiu, Romania
- Novartis Investigative Site, Moscow, Russia
- Novartis Investigative Site, Bratislava, Slovakia
- Spain (3):
  - Novartis Investigative Site, Manresa, Espana
  - Novartis Investigative Site, Barakaldo, Vizcaya
  - Novartis Investigative Site, Las Palmas de Gran Canaria
- Novartis Investigative Site, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2190

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 11 investigative sites in 7 countries.
Pre-assignment Details: There was a screening period of 4 weeks to assess participants eligibility.
Groups:
- Deferasirox FCT 7mg/kg: Deferasirox film-coated tablet 7mg/kg, oral dose daily (starting dose for the first 12 weeks)
- Phlebotomy: Phlebotomy - standard of care
Period: Overall Study
Arm/Group | Deferasirox FCT 7mg/kg | Phlebotomy
Started | 30 | 15
Completed | 22 | 12
Not Completed | 8 | 3
Not completed — Subject/guardian decision | 4 | 3
Not completed — Adverse Event | 3 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deferasirox FCT 7mg/kg | Phlebotomy | Total
Number analyzed (Participants) | 30 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (8.20) | 52.1 (8.13) | 51.8 (8.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 26 | 12 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 30 | 15 | 45

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Achieving Target SF ≤ 100 μg/L for the First Time
Description: Proportion of participants achieving target serum ferritin (SF) ≤ 100 μg/L on or before Month 24. Participants were considered responders if they met response criteria (target SF ≤100 µg/L) on or before Month 24 (Week 104) during the treatment phase. Any participant who discontinued treatment prematurely before meeting such criterion and participants with unknown or missing SF by Month 24 were counted as non-responder.
Time Frame: Up to Month 24
Population: The Full Analysis Set (FAS) comprised all subjects to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Deferasirox FCT 7mg/kg | Phlebotomy
Number analyzed (Participants) | 30 | 15
percentage of participants
  Responder | 40 [22.7 to 59.4] | 80 [51.9 to 95.7]
  Non-Responder | 60 [40.6 to 77.3] | 20 [4.3 to 48.1]

2. Secondary Outcome: Number of Participants With Ocular Treatment Emergent Adverse Events (AEs)
Description: Number of participants with at least one ocular treatment emergent adverse event (new or worsening from baseline).
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of approximately 108 weeks.
Population: The Safety Set (SS) included all subjects who received at least one administration of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox FCT 7mg/kg | Phlebotomy
Number analyzed (Participants) | 30 | 15
Participants
  At least one ocular AE | 9 | 0
  Treatment-related ocular AEs | 2 | 0

3. Secondary Outcome: Number of Participants With Ocular Treatment Emergent Adverse Events (AEs) by Preferred Term
Description: Number of participants with at least one ocular treatment emergent adverse event (new or worsening from baseline). Preferred terms are based on Medical Dictionary of Regulatory Activities (MedDRA) version 26.0.
Time Frame: as for outcome 2
Population: The Safety Set (SS) included all subjects who received at least one administration of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox FCT 7mg/kg | Phlebotomy
Number analyzed (Participants) | 30 | 15
Participants
  Cataract nuclear | 2 | 0
  Glaucoma | 2 | 0
  Blepharitis | 1 | 0
  Cellulitis orbital | 1 | 0
  Dry eye | 1 | 0
  Eye pain | 1 | 0
  Eye ulcer | 1 | 0
  Macular oedema | 1 | 0
  Open angle glaucoma | 1 | 0
  Optic nerve disorder | 1 | 0
  Panophthalmitis | 1 | 0
  Retinal degeneration | 1 | 0
  Retinal haemorrhage | 1 | 0
  Visual acuity reduced | 1 | 0
  Vitreous haemorrhage | 1 | 0

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of participants with treatment emergent AEs (any AE regardless of seriousness), AEs leading to study treatment discontinuation, and SAEs.
Time Frame: as for outcome 2
Population: The Safety Set (SS) included all subjects who received at least one administration of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox FCT 7mg/kg | Phlebotomy
Number analyzed (Participants) | 30 | 15
Participants
  At least one AE | 28 | 12
  At least one SAE | 7 | 0
  AEs leading to discontinuation | 3 | 0

5. Secondary Outcome: Number of Adverse Events in Participants Who Had Study Treatment Interrupted Due to SF ≤ 100 μg/L and Re-initiated Study Treatment When ≥ 300 μg/L
Description: Number of participants with Adverse Events who interrupt deferasirox FCT at least once due to SF level ≤ 100 μg/L and re-initiate therapy at SF level ≥ 300 μg/L.
  There were no participants that re-initiated therapy when reached 300 ug/L.
Time Frame: Up to 24 months
Population: Participants in the Safety Set who had study treatment interrupted due to SF ≤ 100 μg/L and re-initiated study treatment when ≥ 300 μg/L. There were no patients who re-initiated therapy when reached SF 300 μg/L.
Arm/Group | Deferasirox FCT 7mg/kg | Phlebotomy
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Categorical Analysis of logMAR Score Changes From Baseline to Best Post-baseline Changes in One Eye With More Extreme Change
Description: Visual acuity was measured using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart. A letter score was calculated based on the number of letters that could correctly be identified from specified distances. For low luminance and standard acuity measures, visual acuity was described on a logMAR scale for all measures. For including acuity obtained with the ETDRS letter score, the values were converted to a logMAR scale, using the following formula: logMAR = 1.7-0.02*ETDRS score. With this conversion, a difference from baseline of 0.1 logMAR = 5-letter difference in visual acuity, 0.2 logMAR = 10-letter difference, 0.3 logMAR = 15-letter difference, 0.4 logMAR = 20-letter difference, 0.5 logMAR = 25-letter difference and 0.6 logMAR = 30-letter difference. Decrease in logMAR score category from baseline indicates improvement in visual acuity. The best change from baseline amongst all post baseline visit is presented.
Time Frame: Baseline, Weeks 24, 52, 76 and 104.
Population: The Safety Set (SS) included all subjects who received at least one administration of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox FCT 7mg/kg | Phlebotomy
Number analyzed (Participants) | 30 | 15
Participants
  Best change: Decrease <0.1 | 9 | 4
  Best change: Decrease >=0.1 - <0.2 | 9 | 5
  Best change: Decrease >=0.2 - <0.3 | 1 | 0
  Best change: Decrease >=0.3 - <0.6 | 0 | 0
  Best change: Decrease >=0.6 | 1 | 0
  Best change: Decrease Missing baseline assessment | 2 | 0
  Best change: Decrease No decrease from baseline | 8 | 6

7. Secondary Outcome: Categorical Analysis of logMAR Score Changes From Baseline to Worst Post-baseline Changes in One Eye With More Extreme Change
Description: Visual acuity was measured using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart. A letter score was calculated based on the number of letters that could correctly be identified from specified distances. For low luminance and standard acuity measures, visual acuity was described on a logMAR scale for all measures. For including acuity obtained with the ETDRS letter score, the values were converted to a logMAR scale, using the following formula: logMAR = 1.7-0.02*ETDRS score. With this conversion, a difference from baseline of 0.1 logMAR = 5-letter difference in visual acuity, 0.2 logMAR = 10-letter difference, 0.3 logMAR = 15-letter difference, 0.4 logMAR = 20-letter difference, 0.5 logMAR = 25-letter difference and 0.6 logMAR = 30-letter difference. Increase in logMAR score from baseline indicates worsening in visual acuity. The worst change from baseline amongst all post baseline visit is presented.
Time Frame: Baseline, Weeks 24, 52, 76 and 104.
Population: The Safety Set (SS) included all subjects who received at least one administration of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox FCT 7mg/kg | Phlebotomy
Number analyzed (Participants) | 30 | 15
Participants
  Worst change: Increase <0.1 | 11 | 11
  Worst change: Increase >=0.1 - <0.2 | 10 | 2
  Worst change: Increase >=0.2 - <0.3 | 1 | 2
  Worst change: Increase >=0.3 - <0.6 | 3 | 0
  Worst change: Increase >=0.6 | 0 | 0
  Worst change: Increase Missing baseline assessment | 2 | 0
  Worst change: Increase No increase from baseline | 3 | 0

8. Secondary Outcome: Categorical Analysis of Worst Post-baseline Values of Intraocular Pressure in One Eye With More Extreme Change
Description: Intraocular pressure was measured by tonometry. Intraocular pressure values >5 to ≤21 mmHg were considered normal. The worst post-baseline value corresponds to the worst outcome amongst all post baseline visit
Time Frame: Weeks 24, 52, 76 and 104
Population: The Safety Set (SS) included all subjects who received at least one administration of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox FCT 7mg/kg | Phlebotomy
Number analyzed (Participants) | 30 | 15
Participants
  Worst post-baseline value- <=5 mmHg | 0 | 0
  Worst post-baseline value- >5 to <=21 mmHg | 27 | 12
  Worst post-baseline value- >21 to <=30 mmHg | 1 | 3
  Worst post-baseline value- >30 mmHg | 0 | 0
  missing post-baseline assessment | 2 | 0

9. Secondary Outcome: Categorical Analysis of Changes in Intraocular Pressure From Baseline to Best/Worst Post-baseline Changes in One Eye With More Extreme Change
Description: Intraocular pressure was measured by tonometry. A decrease in intraocular pressure from baseline indicated improvement.
Time Frame: Baseline, up to Week 104
Population: The Safety Set (SS) included all subjects who received at least one administration of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox FCT 7mg/kg | Phlebotomy
Number analyzed (Participants) | 30 | 15
Participants
  Increase from baseline >=5 mmHg and <10 mmHg | 4 | 2
  Increase from baseline >=10 mmHg | 0 | 1
  Decrease from baseline >=5 mmHg and <10 mmHg | 6 | 3
  Decrease from baseline >=10 mmHg | 1 | 0
  No change from baseline or min. change (<5 mmHg) | 17 | 9
  Missing post-baseline values | 2 | 0

10. Secondary Outcome: Number of Participants With Slit Lamp Results for Any Evaluation and Worst Eye
Description: Slit lamp examination was used to evaluate lids, cornea, conjunctiva, iris, anterior chamber, aqueous flare, aqueous inflammatory cells and lens. Any post-baseline abnormalities (not present at baseline) in slit lamp examination were assesses by the investigator and classified as insignificant or clinically significant. Number of participants with slit lamp results (normal, insignificant, significant, missing) for any evaluation and worst eye are reported.
Time Frame: Baseline, up to Week 104
Population: The Safety Set (SS) included all subjects who received at least one administration of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox FCT 7mg/kg | Phlebotomy
Number analyzed (Participants) | 30 | 15
Participants
  Baseline: Normal | 12 | 6
  Baseline: Insignificant | 14 | 9
  Baseline: Significant | 2 | 0
  Baseline: Missing | 2 | 0
  Any post-baseline: Normal | 7 | 3
  Any post-baseline: Insignificant | 18 | 12
  Any post-baseline: Significant | 3 | 0
  Any post-baseline: Missing | 2 | 0

11. Secondary Outcome: Number of Participants With an Increase From Baseline of ≥1 and ≥2 in LOCS III Grades
Description: Lens Opacities Classification System III (LOCS III) grading scales include lens opacities defined as nuclear opalescence (NO), nuclear color (NC), cortical (C) cataract and posterior subcapsular (P) cataract with several degrees of extend, i.e. severity. The LOCS III scale for nuclear opalescence and for nuclear color ranges from 0 to 6. The LOCS III scale for cortical cataract and posterior subcapsular cataract opacity ranges from 0 to 5. For all scales, higher values indicate higher opacity, opalescence, or color (range: NO0/NC0/C0/P0 to NO6/NC6/C5/P5).
  Number of participants with an increase from baseline of ≥1 and increase of ≥2 in LOCS III grades is reported.
Time Frame: Baseline, up to Week 104
Population: The Safety Set (SS) included all subjects who received at least one administration of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox FCT 7mg/kg | Phlebotomy
Number analyzed (Participants) | 30 | 15
Participants
  ≥1 grade increase from baseline | 10 | 5
  ≥2 grade increase from baseline | 2 | 0

12. Secondary Outcome: Number of Participants With Fundus Oculi Results for Any Evaluation and Worst Eye
Description: Fundus oculi examination was used to evaluate peripheral retina, macula, optic nerve, and vitreous hemorrhage. Any post-baseline abnormalities (not present at baseline) in fundus oculi examination were assessed by the investigator and classified as insignificant or clinically significant. Number of participants with fundus oculi results (normal, insignificant, significant, missing) for any evaluation and worst eye are reported.
Time Frame: Baseline, up to Week 104
Population: The Safety Set (SS) included all subjects who received at least one administration of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox FCT 7mg/kg | Phlebotomy
Number analyzed (Participants) | 30 | 15
Participants
  Baseline: Normal | 15 | 10
  Baseline: Insignificant | 12 | 5
  Baseline: Significant | 1 | 0
  Baseline: Missing | 2 | 0
  Any post-baseline: Normal | 12 | 10
  Any post-baseline: Insignificant | 14 | 5
  Any post-baseline: Significant | 2 | 0
  Any post-baseline: Missing | 2 | 0

13. Secondary Outcome: Time to Response (TTR)
Description: Time to response (TTR) is defined as the time from the date of randomization to the date of the first time the SF achieved a value ≤ 100 μg/L during the treatment phase. Participants who did not achieve SF ≤ 100 μg/L were censored as follows: at the last serum ferritin assessment date on or before month 24 (week 104), at the day of randomization if a subject does not have any post-baseline serum ferritin value or at the death date. TTR was analyzed using the Kaplan-Meier method.
Time Frame: Up to Month 24
Population: The Full Analysis Set (FAS) comprised all subjects to whom study treatment has been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Deferasirox FCT 7mg/kg | Phlebotomy
Number analyzed (Participants) | 30 | 15
months | NA [19.4 to NA] — Not estimable due to insufficient number of participants with events. | 13.6 [4.0 to 22.1]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of approximately 108 weeks.
Arm/Group | Deferasirox FCT 7mg/kg | Phlebotomy
All-Cause Mortality (participants affected / at risk) | 1/30 | 0/15
Serious Adverse Events (participants affected / at risk) | 7/30 | 0/15
Other Adverse Events (participants affected / at risk) | 23/30 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox FCT 7mg/kg (N=30) | Phlebotomy (N=15)
Nausea (Gastrointestinal disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thoracic outlet syndrome (Nervous system disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox FCT 7mg/kg (N=30) | Phlebotomy (N=15)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Sinus bradycardia (Cardiac disorders) | 1 | 1
Deafness unilateral (Ear and labyrinth disorders) | 1 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 1
Phobic postural vertigo (Ear and labyrinth disorders) | 0 | 1
Cataract nuclear (Eye disorders) | 2 | 0
Glaucoma (Eye disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
Pyrexia (General disorders) | 2 | 0
Vaccination site pain (General disorders) | 0 | 1
Bone abscess (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 2 | 0
Cystitis (Infections and infestations) | 2 | 0
Ear infection (Infections and infestations) | 1 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 2 | 3
Sinusitis (Infections and infestations) | 0 | 1
Suspected COVID-19 (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood cholesterol increased (Investigations) | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 10 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 2 | 0
Blood uric acid increased (Investigations) | 0 | 1
Glycosylated haemoglobin increased (Investigations) | 0 | 1
Vitamin D decreased (Investigations) | 0 | 1
Folate deficiency (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Dizziness (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 4 | 2
Taste disorder (Nervous system disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 3 | 3
Hypotension (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The results should be interpreted with caution due to low number of participants enrolled in both arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/50/NCT03203850/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT03203850/SAP_001.pdf